CLINICAL TRIAL: NCT05977244
Title: Exploring the Effects of Varying Fat:Carbohydrate Diet Permutations on Gastric Emptying and Metabolic Status Using Human Postprandial Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: Taylor's University (Other); National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PD233/18
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Postprandial Lipemia; Postprandial Glycemia; Gastric Emptying
Keywords: meal composition; P/S ratio; macronutrient distribution; glycemic index; glycemia; lipemia; gut hormones; gastric emptying
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HGI+palm olein (Experimental): 1 portion of HGI(high glycemic index) fried rice, fried with palm olein will be served together with 250 milliliter of plain water.
  Interventions: Other: HGI+palm olein
- HGI+soy bean oil (Experimental): 1 portion of HGI (high glycemic index) fried rice, fried with soybean oil will be served together with 250 milliliter of plain water.
  Interventions: Other: HGI+soy bean oil
- LGI+palm olein (Experimental): 1 portion of LGI (low glycemic index) fried rice, fried with palm olein will be served together with 250 milliliter of plain water.
  Interventions: Other: LGI+palm olein
- LGI+soy bean oil (Experimental): 1 portion of LGI (low glycemic index) fried rice, fried with soybean oil will be served together with 250 milliliter of plain water.
  Interventions: Other: LGI+soy bean oil

INTERVENTIONS:
Other: HGI+palm olein — A 5-hour postprandial feeding intervention with 1-weeks washout in between. Blood samples will be collected at 0 hour (baseline) and up to 5 hours after consumption of test meal.
  Arms: HGI+palm olein
Other: LGI+palm olein — A 5-hour postprandial feeding intervention with 1-weeks washout in between. Blood samples will be collected at 0 hour (baseline) and up to 5 hours after consumption of test meal.
  Arms: LGI+palm olein
Other: HGI+soy bean oil — A 5-hour postprandial feeding intervention with 1-weeks washout in between. Blood samples will be collected at 0 hour (baseline) and up to 5 hours after consumption of test meal.
  Arms: HGI+soy bean oil
Other: LGI+soy bean oil — A 5-hour postprandial feeding intervention with 1-weeks washout in between. Blood samples will be collected at 0 hour (baseline) and up to 5 hours after consumption of test meal.
  Arms: LGI+soy bean oil

SUMMARY:
The aim of this clinical trial is to investigate the effects of the meals moderated by fat and carbohydrate (CHO) quality along with varying macronutrient distribution (CHO: fat) on gut physiology and metabolic outcomes using the human postprandial model with healthy subjects.

The main question[s] it aims to answer are:

1. How does meal composition with different polyunsaturated/saturated (P/S) ratio, glycemic index and macronutrient quantity affect lipemia and glycemia?
2. How does meal composition with different P/S ratio, Glycemic index and macronutrient quantity affect gastric emptying?

DETAILED DESCRIPTION:
The study's objectives will be tested via a randomized, crossover study with 16 diet rotations separated by minimum one week washout period. All recruited subjects will be randomly assigned into 2 groups of 7 each namely HGI and LGI with 9 diet rotations within each group. The study design will be a cross-over trial with the same subjects undergoing all arms of the diet rotations. The subjects will be blinded to the test fats used for each rotation. Body weight measurements will be recorded before each postprandial challenge to minimise weight fluctuations between the test rotations.

Study procedures

1. Oral glucose tolerance test (OGTT) Sessions

   Prior and end of the test meal rotations, subjects will undergo oral glucose tolerance test (OGTT) with a glucose reference drink at 2 random sessions without MRI investigation at Taylor's University or Hospital Cancelor Tuanku Muhriz (HCTM), to get an average value for the plasma glucose and insulin standards for each subject. The glucose reference drink composition will be 50g of anhydrous glucose mixed with 250mL of room temperature water. Blood samples will be collected sequentially at 0, 15, 30, 60, 90,120 and 180 minutes.
2. Test meal sessions

During each postprandial test meal rotations, subjects will consume test meals followed by MRI scans at the MRI center at Hospital Cancelor Tuanku Muhriz(HCTM). For scheduled session, Subjects will be advised to refrain from strenuous physical activity, high calorie or fast-food, supplements and coffee intake for 24 hours preceding each postprandial event. Subjects will be at the clinical center at 7:30 and 8:30a.m, following a 12-hour overnight fast. Upon arrival at the centre,subjects will rest for 10min, followed by body weight, blood pressure and self-monitoring of blood glucose (SBMG) measurements. Subsequently, blood samples will be drawn for metabolic investigations as per study objectives. Sequential postprandial MRI scans before and after test meal intake at 0(fasting), 15, 30, 60, 90, 120, 180, 240 and 300 minutes.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects, (n=12-14) without history of chronic disease(s) with body mass index (BMI) between 18.5-25.0 kg/m2 and normal fasting blood glucose status [<5.4 mmol/L] will be enrolled into the study.

Exclusion Criteria:

1. Using pharmacotherapy that interferes with lipid and glucose metabolism or gastrointestinal transit (constipating drugs) or on oral contraceptives (women).
2. Underweight body mass index (BMI): < 18.5 kg/m2
3. With medical history of cardiovascular disease (CVD), Diabetes Mellitus, dyslipidemia and other chronic diseases,
4. acute or chronic gastrointestinal illness
5. If vulnerable to claustrophobia or anxiety
6. Regular alcohol usage
7. On low-calorie diets
8. Smoking

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-05-21 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Lipemia | 0, 15, 30, 60, 90, 120, 180, 240, 300minutes after ingestion of test meals
  To determine the postprandial changes in triacylglyceride (TAG)
Glycemia | 0, 15, 30, 60, 90, 120, 180, 240, 300minutes after ingestion of test meals
  To determine the postprandial changes of glucose

SECONDARY OUTCOMES:
Gastric emptying | 0, 15, 30, 60, 90, 120, 180, 240, 300minutes after ingestion of test meals
  To determine the postprandial changes in half emptying time
Gut hormone | 0, 15, 30, 60, 90, 120, 180, 240, 300minutes after ingestion of test meals
  To determine the postprandial changes of glucose-dependent insulinotropic polypeptide (GIP)

CONTACTS AND LOCATIONS:
Overall Officials: Gowri Nagapan, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No